CLINICAL TRIAL: NCT00596219
Title: Molecular Effects of Short-Term Celecoxib Treatment on Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-147
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: SQUAMOUS CELL CARCINOMA
Keywords: HEAD; NECK; SQUAMOUS; CARCINOMA
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — celecoxib

SUMMARY:
The purpose of this study is to better understand how to use celecoxib, a popular drug widely used for arthritis, for head and neck cancer patients. Some doctors believe that celecoxib may have helpful effects when used for head and neck cancer. Celecoxib has been shown to prevent some cancers in animals. It has also been used to make standard chemotherapy and radiation work better in both animals and humans. However, all of the previous studies focused on tumors outside the head and neck region. To better understand how to use celecoxib for head and neck cancer patients, doctors at MSKCC are studying the effects of the drug on certain chemicals in the body that are thought to be important for cancer treatment.

This study aims to measure how celecoxib affects those chemicals, which can be found in the tumor, blood, and urine of patients with head and neck cancer. Although celecoxib is already used to treat arthritis, this study will be the first to test the drug in head and neck cancer patients.

DETAILED DESCRIPTION:
The selective cyclo-oxygenase 2 (COX-2) inhibitor, celecoxib (Celebrex, Pfizer Inc.), is being investigated as an anticancer agent in chemoprevention and adjuvant therapeutic regimens in many organ systems including the head and neck, lung, colon, breast and bladder. The mechanisms of action are not fully defined and, to date, there are no data regarding the shortterm molecular effects of celecoxib treatment in human tumor tissues. These data are important for understanding the targets and effects of COX-2 inhibitors in cancer.

Specifically, this pilot study seeks to evaluate the feasibility of determining whether celecoxib treatment inhibits COX-2 expression, alters the intratumor eicosanoid profile, and/or suppresses markers of proliferation and growth in human tumor tissues. In addition, this trial aims to evaluate the feasibility of reliably measuring the effects of celecoxib treatment on biomarkers of angiogenesis, prostaglandin metabolism and select growth factors. The study is titled: "Molecular effects of short-term celecoxib treatment on head and neck squamous carcinoma." In this study, 10 patients identified in the Head and Neck Surgical Oncology clinic at MSKCC with untreated squamous cell carcinoma of the oral cavity or oropharynx will be recruited to participate. Participation will not change the standard of cancer care that the patients receive. At the initial office evaluation the tumor will be biopsied. Blood and urine will also be collected. Patients will then take oral celecoxib (400 mg) twice daily starting exactly 5 days prior to staging examination under anesthesia or definitive resection and including the morning of surgery. The tumor will then be re-biopsied at the time of staging examination under anesthesia or surgical resection. Blood and urine will similarly be re-collected at that time.

ELIGIBILITY:
Inclusion Criteria:

* Untreated squamous cell carcinoma of the oral cavity or oropharynx.
* Older than 18 years of age.
* Understand and sign informed consent.

Exclusion Criteria:

* Any prior treatment of the index cancer (chemotherapy, immunotherapy, hormonal therapy or radiation therapy) or similar treatment of an unrelated malignancy within 6 weeks of enrollment into this study.
* Breast-feeding, pregnancy or of childbearing potential (including at least two years post menopause) and unable to confirm adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since last menses.
* History of esophageal, gastric or duodenal ulceration within 6 weeks of enrollment.
* History of acute or chronic renal disorder (blood creatinine level > 1.5 mg/dL).
* History of acute or chronic hepatic disorder or a significant bleeding disorder.
* History of chronic inflammatory disease (e.g. ulcerative colitis, Crohn's disease,rheumatoid arthritis or pancreatitis).
* History of myocardial infarction, angina, or coronary artery disease within the past 6 months, or active cardiac disease.
* The subject is of New York Heart Association (NYHA) Class 3 or 4 cardiac status.
* Corticosteroid use within 6 weeks of enrollment, excluding topical nasal sprays.
* NSAID (including celecoxib) or aspirin (> 81 mg/day) use within 1 week of enrollment.
* History of hypersensitivity to COX-2 inhibitors, NSAIDs, salicylates, or sulfonamides.
* Currently taking fluconazole or lithium.
* Investigational medication use within 6 weeks of enrollment or is scheduled to receive an investigational drug during the course of the study.
* Principal Investigator deems subject to be at high risk for non-compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
• To determine feasibility of measuring molecular changes (COX-2 mRNA, eicosanoid profiles, Ki67, p-EGFR) in head and neck squamous cell carcinoma induced by short-term celecoxib treatment. | 6 years

SECONDARY OUTCOMES:
To evaluate feasibility of measuring effect of short-term celecoxib treatment on blood & urinary concentrations of angiogenesis markers/on blood concentrations of IGF-1 & IGFBP-3/on urinary concentration of PGE-M. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jay Boyle, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org